CLINICAL TRIAL: NCT04891224
Title: Implementation and Evaluation of the Pathway Platform: A Digitally Enabled Care Pathway to Improve Depression Key Performance Indicators and Patient Outcomes in Primary Care Clinics
Brief Title: Use of a Digitally Enabled App With Clinical Team Interface in the Management of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Takeda (Industry); Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9050020
Record Dates: First submitted 2021-03-09; First posted 2021-05-18 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
Keywords: PHQ-9, Shared decision making
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This study will used a pre- post- study design to assess the impact of implementing the Pathway Platform in the primary care setting. Clinic performance and select patient outcomes are compared before and after implementation. Additional patient outcomes are assessed after implementation among patients using the Pathway Platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathway Platform application use (Other): Study participants will download the Pathway app to their mobile device. This app will gather patient health data, present standardized questionnaires and research data collection tools. Subject responses will be visible to their provider via interface with the electronic medical record.
  Interventions: Other: Pathway Platform mobile app

INTERVENTIONS:
Other: Pathway Platform mobile app — The pathway platform intervention involves 3 components: 1. The patient facing app which will: a) Gather health information related to depression management and patient-Provider engagement. b) Clinical data collection; PHQ-9, WHO-5, PDQ-D-5, medication adherence and side effects, goal setting and goal tracking. c) Research data; Patient Activation Measure -13[PAM-13], CollaboRATE, and Work and Social Adjustment Scale [WSAS]. 2. Electronic Medical Record Integration - a) Data collected in the app is accessible to care team in real time. b) Provide a longitudinal summary to assist in decision making and depression management. 3. Educational Scaffolding - a) Training program describing how the Pathway Platform can support care team members in clinical processes related to measurement-based care and shared-decision making. b) Includes ongoing feedback with up to three audit cycles.

SUMMARY:
This study was conducted to understand the use of a mobile app (titled Pathway) to help patients track depression symptoms, medications, side effects, and goals in addition to the usual care with their doctor. Investigators compared the effect of the app over 6 months and examine whether the app can increase engagement between patients and their doctor and help in the management of illnesses as patients started a new treatment for depression. The investigators hoped that using an app to facilitate management of depression symptoms, medication use, and side effects help patients and their providers understand their response to medications and lead to better response and improvements in depression.

DETAILED DESCRIPTION:
A pre- and post- study design was utilized to assess the impact of implementing the Pathway Platform in the primary care setting. The Pathway Platform consists of a mobile app for patients and a care team interface that can be accessed through Epic (electronic medical record system). Eight primary care sites were identified to participate in the study. Care team members involved in depression management received education on evidence-based clinical practices for depression care, such as measurement-based care practices and shared- decision making. Clinics with behavioral resources also received additional education on behavioral health integration. Training on how to onboard patients to use the Pathway Platform and utilize electronic medical records to view data collected in the Pathway Platform was also provided. Study outcomes identified in this protocol are described among patients enrolled in the Pathway Platform (post-implementation cohort) as well as a similar group of patients from the same participating clinics prior to study implantation (pre-implantation cohort). Implementation success was evaluated by comparing study outcomes among these two cohorts. The primary outcome is PHQ-9 utilization over six months are compared between the pre- and post- implementation cohorts. Additional process measures compared include; shared-decision making, medication adjustments, referrals to behavioral health, primary care follow-up post hospitalizations, and depression remission and response. Data collected in the Pathway Platform is also used to explore pre-defined patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with major depressive disorder or reference to "clinical depression" in patient charts.
* Recently prescribed monotherapy antidepressant medication (defined as new start, medication switch, or dose change in the past 3 months.)
* Patients with inadequate response or tolerability concerns determined based on A PHQ-2 score of 3 or greater or a PHQ-9 score of 5 or more, recorded in medical records in the past 6 weeks or during screening,
* Able and willing to provide informed consent
* Able to use the Pathway Platform based on clinician's judgment, e.g. owns an iPhone version 5 or later or smartphones with Android operating systems, have an active data plan or regular WiFi access

Exclusion Criteria:

* Missing PHQ-2 score in the past 6 weeks and/or unable to perform PHQ-2 at index visit
* Diagnosis with bipolar depression, schizophrenia, and/or schizoaffective disorder
* Patient no longer under primary care for depression and has transitioned to a psychiatric care team (i.e., Psychiatrist, Advance Practice Psychiatric Nurse, Psychiatric Nurse Practitioner, Psychiatric Physician Assistant).
* Lack of functional English literacy (indicated by primary language in electronic medical record).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kemp, MD, Principal Investigator — Advocate Medical Group
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lam RW, Lamy FX, Danchenko N, Yarlas A, White MK, Rive B, Saragoussi D. Psychometric validation of the Perceived Deficits Questionnaire-Depression (PDQ-D) instrument in US and UK respondents with major depressive disorder. Neuropsychiatr Dis Treat. 2018 Oct 29;14:2861-2877. doi: 10.2147/NDT.S175188. eCollection 2018. PMID 30464471
- [Background] Krieger T, Zimmermann J, Huffziger S, Ubl B, Diener C, Kuehner C, Grosse Holtforth M. Measuring depression with a well-being index: further evidence for the validity of the WHO Well-Being Index (WHO-5) as a measure of the severity of depression. J Affect Disord. 2014 Mar;156:240-4. doi: 10.1016/j.jad.2013.12.015. Epub 2013 Dec 25. PMID 24412323
- [Background] Chen X, Hu N, Wang Y, Gao X. Validation of a brain-computer interface version of the digit symbol substitution test in healthy subjects. Comput Biol Med. 2020 May;120:103729. doi: 10.1016/j.compbiomed.2020.103729. Epub 2020 Mar 25. PMID 32250858
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] McGahuey CA, Gelenberg AJ, Laukes CA, Moreno FA, Delgado PL, McKnight KM, Manber R. The Arizona Sexual Experience Scale (ASEX): reliability and validity. J Sex Marital Ther. 2000 Jan-Mar;26(1):25-40. doi: 10.1080/009262300278623. PMID 10693114
- [Background] Vortel MA, Adam S, Port-Thompson AV, Friedman JM, Grande SW, Birch PH. Comparing the ability of OPTION(12) and OPTION(5) to assess shared decision-making in genetic counselling. Patient Educ Couns. 2016 Oct;99(10):1717-23. doi: 10.1016/j.pec.2016.03.024. Epub 2016 Mar 24. PMID 27085518
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Forcino RC, Barr PJ, O'Malley AJ, Arend R, Castaldo MG, Ozanne EM, Percac-Lima S, Stults CD, Tai-Seale M, Thompson R, Elwyn G. Using CollaboRATE, a brief patient-reported measure of shared decision making: Results from three clinical settings in the United States. Health Expect. 2018 Feb;21(1):82-89. doi: 10.1111/hex.12588. Epub 2017 Jul 5. PMID 28678426
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Derived] Khatib R, McCue M, Blair C, Roy A, Franco J, Fehnert B, King J, Sarkey S, Chrones L, Martin M, Kabir C, Kemp DE. Design and Implementation of a Digitally Enabled Care Pathway to Improve Management of Depression in a Large Health Care System: Protocol for the Implementation of a Patient Care Platform. JMIR Res Protoc. 2023 Jun 23;12:e43788. doi: 10.2196/43788. PMID 37351941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pathway platform was implemented with interested PCPs from 8 primary care sites.
  Pre- implementation control cohort was created by identifying potentially eligible patients retrospectively from EHR.
  Post-implementation Pathway Cohort - The first participant was enrolled in on 7/21/21 and last participant was enrolled on 7/2/22.
Groups:
- Pre-Implementation Cohort: Retrospective control group identified from study sites.
- Pathway Participants: Consented and activated Pathway app.
Period: Screening
Arm/Group | Pre-Implementation Cohort | Pathway Participants
Started | 90 | 89
Completed | 90 | 89
Not Completed | 0 | 0
Period: Enrollment
Arm/Group | Pre-Implementation Cohort | Pathway Participants
Started | 90 | 89
Completed | 90 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-Implementation Cohort (N=90): Retrospective control group identified from study sites.
- Pathway Participants (N=89): Consented and activated Pathway app.
- Total: Total of all reporting groups
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89) | Total
Number analyzed (Participants) | 90 | 89 | 179
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [28 to 57] | 35 [28 to 46] | 37 [37 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 71 | 123
  Male | 38 | 18 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity , N (%): White | 50 | 41 | 91
  Race/Ethnicity , N (%): Hispanic / Latino | 16 | 16 | 32
  Race/Ethnicity , N (%): Black | 14 | 29 | 43
  Race/Ethnicity , N (%): Other | 10 | 3 | 13
Type of Insurance [Count of Participants; unit: Participants]
  Medicare | 14 | 6 | 20
  Commercial | 59 | 68 | 127
  Medicaid | 17 | 15 | 32
Qualifying PHQ Score [Median (Inter-Quartile Range); unit: units on a scale] — Scores from this nine item questionnaire can range from 0 - 27. Higher scores indicate greater severity of depression.
  units on a scale | 14 [11 to 17] | 15 [12 to 18] | 15 [10 to 18]
Medications at the qualifying visit [Count of Participants; unit: Participants]
  Selective Serotonin Reuptake Inhibitors (SSRIs) | 69 | 67 | 136
  Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs) | 7 | 3 | 10
  Alpha-2 Receptor Antagonists (Tetracyclics ) - Mirtazapine | 2 | 1 | 3
  Tricyclic Agents | 0 | 1 | 1
  Serotonin Modulators | 1 | 0 | 1
  Trintellix | 0 | 0 | 0
  Bupropion | 11 | 17 | 28

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Completed Patient Health Questionnaire
Description: Proportion of patients who have at least 2 Patient Health Questionnaire (PHQ) scores documented in their medical record over the 6 month study period will be compared between pre- and post- Pathway app implementation to determine if there is a change in adherence to measurement based care practices following the implementation of the Pathway Platform in a primary care setting.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Number; unit: participants
Arm/Group | Pre-Implementation Cohort | Pathway Participants
Number analyzed (Participants) | 90 | 89
participants | 35 | 49

2. Secondary Outcome: Process Outcome: Measurement-based Care
Description: The proportion of patients reflecting measurement-based care informed major depression disorder treatment adjustments in their charts, defined as at lease one medication dose change, switch or add on medication.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Number; unit: participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
participants | 38 | 40

3. Secondary Outcome: Process Outcome: Shared-decision Making
Description: The proportion of patients reflecting shared-decision making using the OPTION12 Tool framework.
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway Platform app
Population: Option 12 tool was not utilized in the study because it would have required observation of patient/provider interaction and scoring of the tool by a 3rd party which took place during the pilot study, however was not feasible for this project. Use of this tool required additional research staff to observe in the clinic which we did not have adequate budget to support.
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Process Outcome: Referrals to Behavioral Health
Description: The proportion of patients with at least one referral will be compared.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Number; unit: participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
participants | 21 | 8

5. Secondary Outcome: Process Outcome: Total Number of Hospitalized Participants During Follow up Period
Description: The number who receive follow-up within 7 days of discharge and within 30 days of discharge.
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway Platform app.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
Participants | 19 | 23

6. Secondary Outcome: Process Outcome: Follow-up After Emergency Department Visit for Mental Illness
Description: The proportion of adults who receive follow-up within 7 days of discharge and within 30 days of emergency department visit.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Population: Data for emergency department visits (ED) and ED visits related to behavioral health were analyzed for Pre-implementation cohort and Pathway participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
Participants | 3 | 0

7. Secondary Outcome: Process Outcome: Healthcare Resource Utilization, Hospital Admissions
Description: The number of hospital admissions among patients receiving care at a clinic participating in this study.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Population: Data were analyzed for hospitalization and behavioral health related hospitalizations for both cohorts.
Measure: Number; unit: participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
participants
  Hospitalizations | 19 | 23
  Behavioral health related hospitalization | 4 | 0

8. Secondary Outcome: Process Outcome: Number of Behavioral Related Hospitalizations
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway Platform app.
Population: The data on length of stay for hospitalizations among patients receiving care at a clinic participating in this study was not analyzed because the analytics team was unable to accurately determine and report length of stay (los) for patients in both cohorts. Dates of service were not extracted, unable to provide LOS or time to follow up with primary care physician.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
Participants | 4 | 0

9. Secondary Outcome: Process Outcome: Healthcare Resource Utilization, Emergency Room Admissions
Description: The number of emergency room admissions among patients receiving care at a clinic participating in this study.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
Participants | 11 | 5

10. Secondary Outcome: Process Outcome: Healthcare Resource Utilization, Outpatient Visits
Description: The number of outpatient encounters among patients receiving care at a clinic participating in this study.
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway Platform app.
Population: It was not feasible to accurately gather this information on patients in both cohorts because patients can seek care outside of our healthcare system.
Measure: Number; unit: number of units
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 90 | 89
number of units
  Number of ED Visits | 11 | 5
  Number of Behavioral Health-Related ED Visits | 11 | 5
  Number of Outpatient Visits | 216 | 243

11. Secondary Outcome: Process Outcome: Primary Care Physician (PCP) Visits
Description: The costs associated with health care services among patients receiving care at a clinic participating in this study. Costs will be calculated using USA national average costs for inpatient and outpatient visits.
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway Platform app.
Population: The costs associated with health care services among patients receiving care at a clinic participating in this study was not collected because the study team was not able to obtain financial data. We did not have resources to determine this information or analyze the data as study timeline did not allow. Data will not ever be collected for this outcome.
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Patient Health Questionnaire-9 [PHQ-9] Score
Description: Median Patient Health Questionnaire-9 [PHQ-9] scores <=5 at the end of the study period. Scores from this nine item questionnaire can range from 0-27. Higher scores indicate greater severity of depression. The last measurement available will be used to calculate remission. For participants 'Baseline' refers to the PHQ9 value the patient entered on the day they downloaded the app. For pre-implementation controls 'Baseline' refers to the PHQ value from the EHR on the qualifying visit.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Median (Inter-Quartile Range); unit: median PHQ-9 total score
Arm/Group | Pre-Implementation Cohort | Pathway Participants
Number analyzed (Participants) | 90 | 89
median PHQ-9 total score
  PHQ-9 Median Score: Baseline | 14.5 [11.0 to 27.0] | 12 [9.0 to 17.0]
  3-months | 11.0 [8.5 to 12.5] | 8.5 [3.0 to 15.0]
  6-months | 17.0 [14.5 to 20.0] | 6.5 [3.0 to 12.5]

13. Secondary Outcome: Patient Health Questionnaire-9 [PHQ-9] Score Reduction
Description: Number of patients with a 50 percent or greater reduction in PHQ-9 scores. Scores from this nine item questionnaire can range from 0-27. Higher scores indicate greater severity of depression. A 50 percent reduction in score reflects significant improvement in depression. The first and last scores available during the study period will be used to calculate response.
Time Frame: Baseline to 6 months post-implementation of the Pathway app
Measure: Number; unit: participants
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 7 | 20
participants | 2 | 7

14. Other Pre Specified Outcome: Patient Reported Outcomes: Patient Activation Measure-13 [PAM-13]
Description: This tool consists of 13 statements used to describe one's health. Patients rate each statement on a likert scale from Disagree Strongly (1) to Agree Strongly (4). Sum scores are categorized into levels of activation with higher scores indicating a patient's readiness to take action. The difference between baseline and 6-month follow up will be compared among patients using the Pathway Platform.
Time Frame: Baseline and 6-month post-Pathway app use
Population: Only 54 patients out of the 89 Pathway participants completed a baseline and 6-month Patient Activation Measure-13.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 54
score on a scale | 4 [-5 to 13]

15. Other Pre Specified Outcome: Patient Reported Outcomes: CollaboRATE
Description: CollaboRATE is a process measure of shared decision making between patients and clinicians. Scores from this questionnaire range from 0 -100 with higher scores reflecting more shared decision making. Scores from this tool will be analyzed across 3 time-points.
Time Frame: Baseline, 3 months and 6 months post-Pathway app use.
Population: This tool is intended to be calculated when 3 items have been completed for at least 25 clinical encounters for one particular clinician None of the participants completed this tool at all 3 time-points making the tool invaluable. This outcome only applies to pathway arm.
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Patient Reported Outcomes: Work and Social Adjustment Scale (WSAS)
Description: This tool consists of 5 questions related to a patient's perception of how his/her current problem impairs his/her ability to carry out normal activities. Items are ranked from 0 (not impairing abilities at all) to 8 (very severely impairing abilities). Resulting scores range from 0-40 with higher scores reflecting more severe psychopathology. Baseline and post-Pathway app use scores will be compared among patients using the Pathway Platform.
Time Frame: Baseline and 6-month post-Pathway app use
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 54
score on a scale | -4 [-14 to 6]

17. Other Pre Specified Outcome: Exploratory - Patient Clinical and Reported Outcomes: Patient Health Questionnaire [PHQ-9]
Description: The difference in PHQ-9 scores will be compared in all patients who completed this scale at 2 time points. Scores from this nine item questionnaire can range from 0 - 27. Higher scores indicate greater severity of depression. The difference between two scores and the direction of the change will reflect degree of improvement or decline.
Time Frame: 6 months prior to and 6 months post-implementation of the Pathway app
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pre-Implementation Cohort (N=90) | Pathway Participants (N=89)
Number analyzed (Participants) | 7 | 14
score on a scale | 2 [1 to 3] | 4 [2.5 to 4.5]

18. Other Pre Specified Outcome: Exploratory - Patient Clinical and Reported Outcomes: World Health Organization- Five Well Being Index [WHO-5]
Description: The WHO-5 asks patients to rate 5 indices of wellbeing on a 5 point likert scale; 0 being the worst, 5 being the best. Resulting scores range from 0-25, the higher the score, the better the perceived quality of life. Changes in scores will be compared in patients who completed this scale at 2 time points.
Time Frame: Baseline to 6-month post-Pathway app use
Population: Pre-implementation cohort did not complete these assessments.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 89
score on a scale | 3 [-1 to 7]

19. Other Pre Specified Outcome: Exploratory - Patient Clinical and Reported Outcomes: Perceived Deficits Questionnaire-Depression [PDQ-D5]
Description: The PDQ-5 asks patients to respond to five questions representing four subscales:
  Attention/Concentration, Retrospective Memory, Prospective Memory, and Planning/Organization. Total PDQ-5 score consists of the sum of the raw scores on these 5 items and could range from 0-20 with higher scores indicating greater perceived deficit. The difference in PDQ-D5 scores will be compared in all patients who completed this scale at 2 time points.
Time Frame: Baseline to 6-month post-Pathway app use
Population: Pre-implementation cohort did not complete these assessments.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 89
score on a scale | 4 [0 to 8]

20. Other Pre Specified Outcome: Exploratory - Patient Clinical and Reported Outcomes: Patient Reported Therapeutic Response to Antidepressant Medication Plan.
Description: This Patient Clinical and reported outcome summarizes patient self-reported adherence to antidepressant medication plan as prescribed will be described.
Time Frame: throughout 6-month of Pathway app use
Population: Pre-implementation cohort did not complete these assessments.
Measure: Number; unit: participants
Arm/Group | Pathway Participants (N=89)
Number analyzed (Participants) | 89
participants | 87

ADVERSE EVENTS:
Time Frame: Baseline through week 75
Description: Only data collected prospectively on Pathway cohort is reported here. All spontaneously reported SAEs collected. Causality to study procedures for all SAEs = related/not related to the intervention. AE/SAE/mortality data not collected for retrospective Pre-Implementation Cohort, so it cannot be reported.
Groups:
- Pre-Implementation Cohort Retrospective Control Group Identified From Study Sites.: Retrospective control group identified from study sites.
Arm/Group | Pathway Platform Application Use | Pre-Implementation Cohort Retrospective Control Group Identified From Study Sites.
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/89 | 0/0
Other Adverse Events (participants affected / at risk) | 10/89 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pathway Platform Application Use (N=89) | Pre-Implementation Cohort Retrospective Control Group Identified From Study Sites. (N=0)
Attempted Overdose hospitalization (Psychiatric disorders) | 1 | NA
Hospitalization for Cholecystectomy (Gastrointestinal disorders) | 1 | NA
D & C procedure (Pregnancy, puerperium and perinatal conditions) | 1 | NA
Mitral Valve repair (Cardiac disorders) | 1 | NA
Dizziness (Ear and labyrinth disorders) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pathway Platform Application Use (N=89) | Pre-Implementation Cohort Retrospective Control Group Identified From Study Sites. (N=0)
Carpel tunnel surgery (Musculoskeletal and connective tissue disorders) | 2 | NA
Scar Repair (Surgical and medical procedures) | 1 | NA
L sided chest pain, ED visit (Investigations) | 1 | NA
Abdominal pain/Ovarian cyst rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Observational hospitalization for abnormal vaginal bleeding (Reproductive system and breast disorders) | 1 | NA
L Breast Mass Excision (Reproductive system and breast disorders) | 1 | NA
Laparoscopic Lysis of Adhesions (renal) (Surgical and medical procedures) | 1 | NA
ED visit Anxiety (General disorders) | 1 | NA
ED Visit Cellulitis R hand (Skin and subcutaneous tissue disorders) | 1 | NA

LIMITATIONS AND CAVEATS:
Small sample size and high attrition rates in both cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04891224/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04891224/ICF_001.pdf